CLINICAL TRIAL: NCT04526002
Title: The Utility of Concurrent TBS/fNIRS for Antidepressant Treatment Optimization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Georg Kranz (Other)
Collaborators: Chinese University of Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Kowloon Hospital, Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15100120
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Theta-Burst Stimulation; Major depression; Treatment prediction; Functional NIRS; Concurrent TBS/fNIRS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients with MDD and healthy controls will undergo TBS/fNIRS to investigate the direct effects of TBS of healthy and presumed neuropathological prefrontal cortex.
  This is followed by a 4-week TBS treatment for MDD patients in order to evaluate the relationship between immediate excitability modulations of the DLPFC and treatment response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Concurrent TBS/fNIRS with iTBS and followed by cTBS after 1h (Experimental): self-explanatory, see Arm Title
  Interventions: Device: Theta-burst stimulation (TBS)

INTERVENTIONS:
Device: Theta-burst stimulation (TBS) — TBS comprises 3-pulse 50-Hz bursts, applied every 200 ms (at 5 Hz) as described previously (Huang, Edwards et al. 2005). iTBS consists of 2-second trains with an inter-train-interval of 8 seconds. We will repeat trains (30 pulses; 10 bursts) for 20 times to reach a total number of 600 pulses (3x10x20). cTBS will comprise uninterrupted bursts to reach a total number of 600 pulses, as done routinely by others. Concurrent TBS/fNIRS stimulation will be applied over the left (iTBS) and right (cTBS) DLPFC at an intensity of 70-120%* resting motor threshold (RMT) (The ideal %RMT will be determined first in a pilot study). In part two, stimulation intensity for patients will be 120% RMT (titration to full therapeutic dose over the first three days), as approved by the FDA in the U.S. (Blumbeger et al. 2018). The stimulation site will be the same as in the concurrent TBS/fNIRS stimulation (see above).
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) with theta bursts (i.e. TBS) of the dorsolateral prefrontal cortex (DLPFC) is an innovative treatment for major depressive disorder (MDD). Indeed, the U. S. Food and Drug Administration (FDA) has only recently approved TBS (in August 2018). However, fewer than 50% of patients show sufficient response to this treatment; markers for response prediction are urgently needed. Moreover, there is a lack of knowledge of the mechanism of action of TBS of the DLPFC. This is due to difficulties of directly measuring prefrontal stimulation effects, as compared to the stimulation of motor cortex and utilizing motor evoked potentials as direct readout. However, knowledge of immediate DLPFC modulation by TBS is necessary to extrapolate downstream effects on the neural and symptoms level.

Thus, there is a need for research that aims to quantify the direct and immediate after-effects of TBS on DLPFC function. Most importantly, with regard to precision medicine, there is a need for research that explores the utility of immediate DLPFC reactivity to TBS for the prediction of antidepressant treatment response. There is common agreement that certain forms of rTMS inhibit or excite brain activity, respectively. However, evidence indicates that there is considerable individual variability in the brain responses to rTMS. Whether differences in individual DLPFC modulation by rTMS can be utilized as a predictive marker for treatment response remains to be investigated.

This research program will exploit the combination of functional near-infrared spectroscopy (fNIRS) with brain stimulation. Concurrent TBS/fNIRS measurements will allow us to systematically investigate TBS-induced modulation of blood oxygenation as a proxy for induced brain activity changes. The findings from this study will (1) elucidate the immediate effects of excitatory and inhibitory TBS on prefrontal activity in TBS treatment-naïve patients with MDD and (2) validate the potential utility of TBS-induced brain modulation at baseline for the prediction of antidepressant response to four weeks of daily TBS treatment.

Major depression is a severe mental disorder and is associated with considerable economic costs but adequate treatments are poorly explored. This research program will pave the way towards an affordable and easy-to-implement method for response prediction before treatment commencement. Thus, our research proposal has high potential to inform tailored treatment strategies, as envisaged in precision medicine.

DETAILED DESCRIPTION:
Please refer to the full proposal

ELIGIBILITY:
MDD group:

Inclusion Criteria:

* MDD (DSM-5), HAMD17 ≥18, approval for TBS treatment by the physician in charge, stable antidepressive medication 4 weeks before treatment (the sample will include at least 20 drug-naïve patients in order to avoid confounding effects of medication for testing hypothesis 4).

Exclusion Criteria:

* a history of brain surgery, head injury, stroke or neurodegenerative disorder, diagnosis of personality disorder, psychotic features, active suicidal intent, severe somatic comorbidities, cardiac pacemakers, deep brain stimulation, intracranial metallic particles, history of seizures, antiepileptics and benzodiazepines corresponding to a dose of >1 mg lorazepam/d, substance dependence or abuse, if it is the primary clinical problem.

HC group:

Inclusion Criteria:

* age between 18 and 60, right-handedness.

Exclusion Criteria:

* a current or previous diagnosis of a psychiatric, neurological disorder or severe internal illness, common contraindications to rTMS,26 and a psychiatric disorder in their first-degree relatives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Response rate after treatment (Montgomery-Asberg depression rating scale, MADRS reduction ≥50% of baseline) | post treatment, up to 22 months
  We will use the MADRS as the primary outcome measure because this symptom rating scale is more sensitive to changes over time. The score of MADRS is ranging from 0 to 60, with higher scores indicative of greater depressive symptomology.
Oxygenated hemoglobin (HbO) change compared to baseline | during and post TBS-fNIRS measurement, an average of 2 months. As well as at follow-up, up to 30 months
  TBS-induced HbO change in the DLPFC during and after stimulation

SECONDARY OUTCOMES:
Remission rate after treatment (MADRS≤10) | post treatment, up to 22 months
  See above
Absolute change of mean Hamilton depression rating scale (HAMD17) after 2 and 4 weeks of treatment, as well as at 1 month follow-up | at follow-up, up to 30 months
  The score of HAMD is ranging from 0 to 53, on which increasing scores represent increasing severity of symptoms
Absolute change of mean Inventory of depression symptomatology-clinician (IDS-C30) after 2 and 4 weeks of treatment, as well as at 1 month follow-up | at follow-up, up to 30 months
  The score of IDS-C30 ranges from 0 to 84, on which increasing scores represent increasing severity of symptoms
Hb change compared to baseline | during and post TBS-fNIRS measurement, an average of 2 months. As well as at follow-up, up to 30 months
  TBS-induced Hb change in the DLPFC during and after stimulation
the area under curve of HbO and Hb value during stimulation | during TBS-fNIRS measurement, an average of 2 months. As well as at follow-up, up to 30 months
  TBS-induced HbO and Hb change in the DLPFC during stimulation
the steepness of the Hb and HbO values change | during TBS-fNIRS measurement, an average of 2 months. As well as at follow-up, up to 30 months
  TBS-induced HbO and Hb change in the DLPFC during stimulation

OTHER OUTCOMES:
Change of Patient Health Questionnaire (PHQ-9, Chinese version) at each treatment day | till to end of treatment, up to 18 months
  The score of PHQ-9 ranges from 0 to 27, on which increasing scores represent increasing severity of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kan RLD, Mak ADP, Chan SKW, Zhang BBB, Fong KNK, Kranz GS. Protocol for a prospective open-label clinical trial to investigate the utility of concurrent TBS/fNIRS for antidepressant treatment optimisation. BMJ Open. 2022 Feb 10;12(2):e053896. doi: 10.1136/bmjopen-2021-053896. PMID 35144953